CLINICAL TRIAL: NCT01033955
Title: Collaborative H1N1 Adjuvant Treatment (CHAT) Pilot Trial
Brief Title: Collaborative H1N1 Adjuvant Treatment Pilot Trial
Acronym: CHAT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: H1N1 pandemic concluded in early 2010
Sponsor: Canadian Critical Care Trials Group (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Physicians' Services Incorporated Foundation (Other); Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 001 CHAT 2009
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Critically Ill; H1N1/Influenza Infection
Keywords: critical care; H1N1/influenza infection; respiration; ventilation, artificial; critically ill patients; invasive mechanical ventilation; H1N1/influenza infection (suspected, probable or confirmed)
MeSH Terms: conditions — Critical Illness; Respiratory Aspiration | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug (Rosuvastatin) Crestor (Experimental): The first dose of encapsulated study drug or placebo (day 1) will be administered within 4 hours of randomization as a loading dose of 40 mg. The placebo will be identical in appearance to Rosuvastatin. Thereafter, doses of 20 mg will be administered daily starting on the next calendar day at 10 pm daily (+/- 4 hours) as a maintenance dose from days 2 to 14. If the patient is of Asian descent, is <18 years, or serum creatinine is greater than or equal to 248 μmol/L (2.8 mg/dL) dose adjustments will be made according to a dose adjustment algorithm.
  Interventions: Drug: Rosuvastatin
- Placebo (Placebo Comparator): An identical appearing placebo will be administered to patients in the second study arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin — Loading dose: 40 mg (day 1) Maintenance dose: 20 mg (days 2-14)
  Other Names: Crestor
  Arms: Drug (Rosuvastatin) Crestor
Drug: Placebo — identical appearing encapsulated placebo.
  Arms: Placebo

SUMMARY:
Study Design: A, multinational, double blind, placebo-controlled pilot RCT involving 80 patients in the general ICUs of 30 centres. Most patients will be recruited from within Canada; however cases will be recruited from international sites. This study will be conducted under the auspices of the Canadian Critical Care Trials Group (CCCTG) and the International Forum for Acute Care Trialists (InFACT).

DETAILED DESCRIPTION:
Primary Objective: The primary objective of the CHAT Pilot Trial is to assess our ability to recruit the desired patient population (i.e., the proportion of eligible patients enrolled in the trial), and to conduct a scientifically rigorous international RCT under pandemic circumstances.

Secondary Objectives: To evaluate (i) adherence to the medication administration regimen. (ii) the ability for research staff to collect the required primary and secondary endpoints for the planned full CHAT trial, (iii) the number of study withdrawals due to administration of open-label statins and withdrawals of consent and (iv) the impact of the approved consent model on recruitment rates.

Study Methods (Overview): Using a web-based randomization system patients, research coordinators will assign critically ill adults treated with antiviral medication for < or equal to 72 hours and requiring mechanical ventilation to one of two treatment strategies (rosuvastatin or placebo) for 14 days. Given the need to recruit patients into the CHAT Trial under pandemic conditions, when family members may not be present to provide written informed consent, we will request either a waiver of consent or deferred consent from Research Ethics Boards (REBs) at participating centres. The Keenan Research Centre/Li Ka Shing Knowledge Institute (St Michael's Hospital, Toronto, Ontario) will be the study Methods Centre.

ELIGIBILITY:
Inclusion Criteria:

1. Critically ill adult patients > or equal to 16 years of age admitted to an adult ICU for any reason with suspected, probable or confirmed influenza infection
2. Requiring mechanical ventilation (invasive or non-invasive)
3. Receiving antiviral therapy (any medication at any dose and for any intended duration) for < or equal to 72 hours
4. Attending physician or intensivist must have a 'moderate' to 'high' index of suspicion for influenza

Exclusion Criteria:

1. Age < 16 years
2. Do not resuscitate or re-intubate order documented on chart or anticipated withdrawal of life support
3. Weight < 40 kg
4. Unable to receive or unlikely to absorb enteral study drug (e.g. incomplete or complete bowel obstruction, intestinal ischemia, infarction, short bowel syndrome)
5. Rosuvastatin specific exclusions:

   * Already receiving a statin (Atorvastatin, Lovastatin, Simvastatin, Pravastatin, Rosuvastatin)
   * Allergy or intolerance to statins
   * Receiving niacin, fenofibrate, cyclosporine, gemfibrozil, lopinavir, ritonavir or planned use of oral contraceptives or estrogen therapy during the ICU stay
   * CK exceeds 10 times ULN or ALT exceeds 8 times the ULN
6. Severe chronic liver disease (Child-Pugh Score 11-15)
7. Previous enrollment in this trial
8. Pregnancy or breast feeding
9. At the time of enrollment, patients must not have received >72 hours of antiviral therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Proportion of eligible patients enrolled in the CHAT Pilot Trial. | anticipated 6 months (duration of pandemic)

SECONDARY OUTCOMES:
Adherence to the medication regimen as outlined in the study protocol. | 14 day treatment course
Proportion of completed primary and secondary endpoints collected for the planned full CHAT trial | 90 days
The number of study withdrawals due to administration of open label statins and consent withdrawals | anticipated 6 month study period

CONTACTS AND LOCATIONS:
Overall Officials: John C Marshall, MD, FRCPS, Principal Investigator — Unity Health Toronto; Karen EA Burns, MD,FRCPC,MSc, Principal Investigator — Unity Health Toronto
Locations (9):
- Canada (9):
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Health Sciences Centre, Winnipeg, Manitoba
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Hopital Laval, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec